CLINICAL TRIAL: NCT03203278
Title: Web-based Exercise Intervention for South Asian People With Type 2 Diabetes: a Randomised Controlled Trial
Brief Title: Web-based Exercise for South Asian People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN17DI329
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: South Asian
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based exercise programme (Experimental): Personalised exercise programme, undertaken three times a week (with no more than two rest days between sessions) for 12 weeks
  Interventions: Behavioral: Web-based exercise programme
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Web-based exercise programme — Aerobic, resistance and balance exercises
  Arms: Web-based exercise programme

SUMMARY:
This randomised controlled trial aims to investigate the effect of a 12 week personalised exercise programme delivered using a web-based platform, compared to usual care, on glycaemic control, muscle strength, functional ability, blood lipid profile, blood pressure and quality of life in adult South Asians with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
A mixed method approach involving both qualitative and quantitative methods will be used.

The quantitative component will consist of a single blind, randomised controlled trial (RCT), which will explore the effects of the intervention on glycaemic control (blood sugar levels) and other secondary outcomes.

The qualitative component will consist of face to face interviews to explore the views of participants regarding acceptability and barriers affecting adherence to this intervention.

Potential participants will be informed about the study at hospital diabetes clinics, community health organisations, support groups, places of worship and General Practitioner (GP) surgeries. Recruitment is estimated to last for 9 months. Potential participants will be sent a participant information sheet (PIS) in either English or Urdu, depending on their preference. Those wishing to take part will meet the researcher at a convenient location, for eligibility screening and consent. If necessary, translation services can be arranged for those with limited English throughout the study.

Following baseline assessment, participants will be randomised to either the intervention or control group. Participants in the control group will be asked to continue their usual care and day to day physical activity routine. In addition, they will be given general information about diabetes management. Participants who wish to use the website for exercise will be provided with access at the end of all assessments.

Participants assigned to the intervention group will be asked to perform a personalised exercise programme, undertaken three times a week (with no more than two rest days between sessions) for 12 weeks. Participants will meet the researcher face to face immediately after randomisation. During this meeting, a brief physical assessment will be undertaken and exercise goals will be discussed and agreed with participants. The researcher will then design a personalised exercise programme for each participant using the resources available on the web-based exercise website. The exercise programme prescription and progression will be in line with American Diabetes Association (ADA) and American College of Sports Medicine (ACSM) guidelines (Colberg et al. 2016). The website (www.webbasedphysio.com) will be used to deliver the intervention. This website has been modified, in collaboration with South Asians, to be culturally suitable for people of South Asian backgrounds in terms of content and language (Albalawi et al, under review). The researcher will contact participants every two weeks via telephone to encourage use of the website, ask about progress, and to deal with any technical issues that they might face while using the website. Participants will be advised to contact the researcher to request a change in their programme or if a problem arises. The researcher will make changes remotely and participants will be informed of any changes by phone or email. Participants will be asked to meet the researcher face to face to discuss progression and goals at week 6 (midway). Regardless of groups allocation, all participants will be assessed three times by a blind assessor at baseline (week=0) , after the end of the intervention (week=12) and 8 weeks after the end of the intervention (week=20).

Assessment of outcome measures will take place at convenient locations and each visit should take no more than 90 minutes. Travel expenses will be provided.

All participants will be informed that they are free to withdraw from the study at any time without being obliged to give notice or provide any explanation. Any data collected before their withdrawal will be considered in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* define themselves as South Asians
* BMI 21 - 29.9 kg/m2
* diagnosed with Type 2 Diabetes Mellitus (T2DM) by a physician more than 6 months previously
* access to a personal computer/tablet, smart phone or smart television with an email address and Internet connection
* able to understand English or Urdu

Exclusion Criteria:

* type 1 diabetes
* any medical conditions that would affect adherence or contraindicate exercise including severe peripheral neuropathy, severe autonomic neuropathy, severe physical limitations, heart disease, pre-proliferative or proliferative retinopathy, uncontrolled hypertension (>180/ 100mmHg), or coronary artery disease.
* people using insulin if they do not have a self-monitoring glucose device or are unable to use such devices.
* engaging in exercise training of 150 minutes a week or more
* participating in other interventional studies aiming to improve glycaemic control
* unwilling to be randomised

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | Baseline to 12 weeks
  Change in HbA1c

SECONDARY OUTCOMES:
Blood lipid profile (cholesterol) | Baseline to 12 weeks
  Change in total cholesterol level
Blood lipid profile (cholesterol) | 12 weeks to 20 weeks
  Change in total cholesterol level
Blood lipid profile (high density lipoproteins) | Baseline to 12 weeks
  Change in high density lipoprotein (HDL) level
Blood lipid profile (high density lipoproteins) | 12 weeks to 20 weeks
  Change in high density lipoprotein (HDL) level
Blood lipid profile (low-density lipoproteins) | Baseline to 12 weeks
  Change in low density lipoprotein (LDL) level
Blood lipid profile (low-density lipoproteins) | 12 weeks to 20 weeks
  Change in low density lipoprotein (LDL) level
Blood lipid profile (triglyceride) | Baseline to 12 weeks
  Change in triglyceride level
Blood lipid profile (triglyceride) | 12 weeks to 20 weeks
  Change in triglyceride level
Blood pressure | Baseline to 12 weeks
  Change in blood pressure result
Blood pressure | 12 weeks to 20 weeks
  Change in blood pressure result
Body mass index (BMI) | Baseline to 12 weeks
  Change in BMI
Body mass index (BMI) | 12 weeks to 20 weeks
  Change in BMI
Waist circumference | Baseline to 12 weeks
  Change in waist circumference
Waist circumference | 12 weeks to 20 weeks
  Change in waist circumference
Ten metre walking test (10MWT) | Baseline to 12 weeks
  Change in 10 MWT result
Ten metre walking test (10MWT) | 12 weeks to 20 weeks
  Change in 10 MWT result
Timed Up and Go test | Baseline to 12 weeks
  Change in Timed Up and Go test result
Timed Up and Go test | 12 weeks to 20 weeks
  Change in Timed Up and Go test result
Muscle power | Baseline to 12 weeks
  Change in hand grip dynamometer score
Muscle power | 12 weeks to 20 weeks
  Change in hand grip dynamometer score
Quality of Life - WHO-QOL BREF score | Baseline to 12 weeks
  Change in World Health Organisation Quality of Life (WHO-QOL BREF) score
Quality of Life - WHO-QOL BREF score | 12 weeks to 20 weeks
  Change in World Health Organisation Quality of Life (WHO-QOL BREF) score
Adherence - exercise diary completion | 12 weeks
  Number of times exercise diary completed
Dietary intake | Baseline to 12 weeks
  Change in Food Frequency Questionnaire score
Dietary intake | 12 weeks to 20 weeks
  Change in Food Frequency Questionnaire score
Change in Medication | Baseline to 12 weeks
  Change in medication
Change in Medication | 12 weeks to 20 weeks
  Change in medication
Glycaemic control | 12 weeks to 20 weeks
  Change in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PhD, Study Director — Glasgow Caledonian University
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No